CLINICAL TRIAL: NCT05887752
Title: Efficacy of Combined Treatment With Hunova® Instrumentation and Standard Rehabilitation, Compared to Standard Rehabilitation, on the Improvement of Trunk Control in Spinal Cord Injured Patients: Hunova® Randomized Controlled Trial
Brief Title: Hunova® Randomized Controlled Trial for Trunk Control Improvement in Spinal Cord Injured Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montecatone Rehabilitation Institute S.p.A. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CE AVEC 286-2023-DISP-AUSLIM; MRI_47-2023 (Other: Montecatone Rehabilitation Institute S.p.A.)
Record Dates: First submitted 2023-05-24; First posted 2023-06-05 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Spinal Cord Injury
Keywords: Robotic rehabilitation; Trunk control; Hunova
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial (add-on in the first half of the study period)
Who Masked: Outcomes Assessor
Masking Description: After selection and enrollment, just before the beginning of the 4-week rehabilitation period, baseline assessments are carried out and patients are randomized. Due to the nature of the Hunova® treatment, blinding of patients and researchers involved in treatment administration will not be possible. Blinding is thus forecast for outcomes' assessors and statisticians only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard rehab plus 20-session Hunova rehabilitation (Experimental): Patients will receive the Standard rehabilitation for a period of 4 weeks.
  In the same 4 weeks and days, the Hunova® rehabilitation (20 sessions in total) will also be administered.
  Interventions: Other: Standard rehabilitation; Device: Hunova® rehabilitation
- Standard rehab plus 10-session, delayed, Hunova rehabilitation (Other): Patients will receive the Standard rehabilitation for a period of 4 weeks.
  During the last 2 weeks, in the same days, the Hunova® rehabilitation (10 sessions in total) will be also administered.
  Interventions: Other: Standard rehabilitation; Device: Hunova® rehabilitation

INTERVENTIONS:
Other: Standard rehabilitation — Carried out 3h/day, 5 days/week at the Montecatone Institute. It implies a multiprofessional approach through:
  * physiotherapy;
  * occupational therapy;
  * sports rehabilitation.
Device: Hunova® rehabilitation — Performed in a dedicated gym of the Montecatone Institute, 1 hour/day, 5 days/week, in the presence of a physiotherapist. Depending on the improvement of the person and of his skills acquisition, the degree of tilting of the Hunova® seat in the various planes may vary.

SUMMARY:
In patients with Spinal Cord Injury (SCI), trunk and therefore postural control (both in statics and dynamics) are impaired, often with strong consequences on daily life activities. Therefore, improvement and reinforcement of trunk control are primary rehabilitation (rehab) goals.

For the evaluation of trunk control in SCI people, still today no tests and scales are definable as gold standards.

Nowadays, for evaluation and rehab purposes of trunk control, balance and proprioception, in both sitting and standing positions, conventional rehabilitation can be supplemented with robotic treatments, e.g. through the Hunova® device (by Movendo Technology). Several studies have demonstrated that conventional rehab associated with robotic training is able to influence functional and motor outcomes in stroke patients, while little evidence is available on SCI patients, also on the number of robotic sessions needed.

The present randomized controlled study primarily aims to demonstrate the effects on trunk control of an integrated rehab treatment (standard plus Hunova®), compared to the standard alone and to gain evidence on the better rehabilitation scheme in terms of number of Hunova® sessions. The correlation between the variation of trunk control, measured by the output data of the Hunova® device itself - ideally more objective - and that assessed through a validated clinical scale, will also be estimated.

DETAILED DESCRIPTION:
In SCI patients trunk and therefore postural control (both in statics and dynamics) are impaired, often with strong consequences on daily life activities. Postural control is defined as the ability to maintain balance despite internal and external perturbations, with the aim of bringing the person's barycenter within his standing area.

Therefore, improvement and reinforcement of trunk control are primary rehab goals.

For the evaluation of trunk control in SCI people, still today no tests and scales are definable as gold standards. Only a few are considered as more reliable, some of them suitable for acute/subacute SCI, some others for chronic SCI. In some published studies, inertial sensors have been used for a more precise evaluation of the Center of Pressure (COP), of the sway area, in relation to the trunk control, but further validation studies are needed. The use of more objective tools could provide additional information on the behavior of SCI people on postural control, thus not only on muscle strength. Of particular interest are the less or more complex compensation strategies implemented and the muscle activation patterns involved in trunk control, assessable through e.g. surface electromyography.

Nowadays, for rehab purposes of trunk control, balance and proprioception, in both sitting and standing position, conventional rehab can be supplemented with robotic treatments, e.g. through the Hunova® device (by Movendo Technology). Several studies have demonstrated that conventional rehab associated with robotic training is able to influence functional and motor outcomes in stroke patients, while little evidence is available on SCI patients, also on the number of robotic sessions needed. The same Hunova® device also allows parameters evaluation by means of its output data.

The present randomized controlled study primarily aims to demonstrate the effects on trunk control of an integrated rehab treatment (standard plus Hunova®), compared to the standard alone and to gain evidence on the better rehab scheme in terms of number of Hunova® sessions. The correlation between the variation of trunk control, measured by the output data of the Hunova® device itself - ideally more objective - and that assessed through a validated clinical scale, will also be estimated.

Randomization will be stratified, based on SCI lesion completeness. A 1:1 allocation ratio will be used for each stratum.

ELIGIBILITY:
Inclusion Criteria:

* Spinal Cord Injury of any etiology;
* American Spinal Injury (AIS) grade A or B and American Spinal Injury Association (ASIA) neurological level T1 or below; alternatively AIS grade C or D and ASIA neurological level C4 or below;
* stable clinical conditions;
* maximum distance from the SCI event: 6 months;
* ability to maintain a sitting position for at least 1h continuously;
* subjects capable and collaborating, able to give in person their informed consent.

Exclusion Criteria:

* wearer of tracheal cannula, with the need for bronchoaspiration;
* wearer of spine orthosis;
* instability or significant deformity of the spine and/or of the lower limbs;
* presence of paraosteoarthropathy (POA) in development/inflammatory phase;
* presence of ischial Pressure Lesion (PL) of stage ≥ 3, according to the National Pressure Ulcer Advisory Panel / European Pressure Ulcer Advisory Panel (NPUAP/EPUAP) classification;
* need for a lifter for patient transfer;
* body weight ≥ 150 kg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change of trunk control after 10 sessions of Hunova® rehabilitation | Baseline (initial assessment); 2 weeks after Baseline
  Evaluation of the efficacy of Hunova® rehabilitation for 10 consecutive sessions (2 weeks treatment period), in addition to the Standard rehab treatment, compared to the Standard treatment only, in terms of improvement of trunk control (both in statics and dynamics), while seated. The validated Trunk Control Test clinical measurement scale for SCI people (TCT-SCI) is employed
Change of trunk equilibrium after 10 sessions of Hunova® rehabilitation | Baseline (initial assessment); 2 weeks after Baseline
  Evaluation of the efficacy of Hunova® rehabilitation for 10 consecutive sessions (2 weeks treatment period), in addition to the Standard rehab treatment, compared to the Standard treatment only, in terms of ability to adapt to external postural perturbations. The validated Trunk Control Test clinical measurement scale for SCI people (TCT-SCI) is employed

SECONDARY OUTCOMES:
Change of trunk control after 20 versus 10 Hunova® rehab sessions | Baseline (initial assessment); 2 weeks after Baseline; 4 weeks after Baseline
  Evaluation of the efficacy of Hunova® treatment for a prolonged period of 20 sessions (4 weeks), compared to a basic treatment of 10 sessions (2 weeks), in terms of improvement of trunk control (both in statics and dynamics), while seated. The validated TCT-SCI scale is employed for assessments
Change of trunk equilibrium after 20 versus 10 Hunova® rehabilitation sessions | Baseline (initial assessment); 2 weeks after Baseline; 4 weeks after Baseline
  Evaluation of the efficacy of Hunova® treatment for a prolonged period of 20 sessions (4 weeks), compared to a basic treatment of 10 sessions (2 weeks), in terms of improvement of ability to adapt to postural perturbations. The validated TCT-SCI scale is employed for assessments
Comparison between trunk control measurements obtained by Hunova® and a validated clinical scale | Baseline (initial assessment); 2 weeks after Baseline; 4 weeks after Baseline
  Estimation, during and after the rehabilitation period, of the correlation between measures of trunk control improvement, given by the Hunova® device itself, and operator-dependent measures obtained through a validated clinical scale (TCT-SCI)
Estimation of correlation between change of trunk control and functional activities - self care | Baseline (initial assessment); 2 weeks after Baseline; 4 weeks after Baseline
  Estimation, during and after the rehabilitation period, of the correlation between improved trunk control (measured by the TCT-SCI scale) and the improvement in functional activities (measured through the Spinal Cord Independence Measure (SCIM) scale, version III, section "Self-care")
Estimation of correlation between change of trunk control and functional activities - overall mobility | Baseline (initial assessment); 2 weeks after Baseline; 4 weeks after Baseline
  Estimation, during and after the rehabilitation period, of the correlation between improved trunk control (measured by the TCT-SCI scale) and the improvement in functional activities (measured by a physician through the Spinal Cord Independence Measure (SCIM) scale, version III, section "Overall mobility");
Estimation of correlation between change of trunk control and patients' self-perception of performances in functional activities | Baseline (initial assessment); 2 weeks after Baseline; 4 weeks after Baseline
  Estimation, during and after the rehabilitation period, of the correlation between the change of trunk control (measured by the TCT scale) and the change of patient's self-perception of the performance (measured by the Canadian Occupational Performance Measure questionnaire - COPM) of those functional activities self-perceived as relevant
Estimation of correlation between change of trunk control and patients' satisfaction with performances in functional activities | Baseline (initial assessment); 2 weeks after Baseline; 4 weeks after Baseline
  Estimation, during and after the rehabilitation period, of the correlation between the change of trunk control (measured by the TCT scale) and the change of patients' satisfaction with the performance (measured by the Canadian Occupational Performance Measure questionnaire - COPM) of those functional activities self-perceived as relevant
Estimation of correlation between change of trunk control and patients' quality of life | Baseline (initial assessment); 2 weeks after Baseline; 4 weeks after Baseline
  Estimation, during and after the rehabilitation period, of the correlation between the change of trunk control (measured by the TCT scale) and the change of quality of life perceived by the study subjects (measured by the questionnaire developed by the World Health Organization of the Quality of Life assessment, shorter version - WHOQOL-BREF)
Change of the COP area as a function of SCI neurologic categories | Baseline (initial assessment); 2 weeks after Baseline; 4 weeks after Baseline
  Analysis of the variation of the Centre Of Pressure (COP) area during and after the rehabilitation period, stratified by the following SCI categories: complete paraplegia with high thoracic SCI (neurological level ≥T6), complete paraplegia with low thoracic SCI (neurological level <T6), incomplete paraplegia and tetraplegia. Measurements will be carried out in centimeters
Change of activity patterns in muscles involved in trunk control, assessed by electromyography | Baseline (initial assessment); 4 weeks after Baseline
  Evaluation of the variation of muscle activity patterns of the muscles contributing to the maintaining of trunk control (latissimus dorsi, trapezius, latissimus pectoralis, erector spinae), between the beginning and the end of the 4-week rehab period under study. Measurements will be carried out through surface dynamic electromyography
Tolerability of the Hunova® rehab treatment | For intervention arm: 2 weeks after Baseline; 4 weeks after Baseline. For comparator arm: 4 weeks after Baseline
  Self-patient's perception of the fatigue during the treatment with Hunova®, associated with the Standard rehabilitation treatment, for trunk control. Assessments are carried out through an in-house developed, self-administered questionnaire at the end of the 4-week rehab period under study
Satisfaction of the Hunova® rehab treatment | Time Frame: 4 weeks after Baseline
  Patient's satisfaction with the Hunova® treatment associated with the Standard rehabilitation treatment for trunk control. Assessments are carried out through an in-house developed questionnaire, administered by a physiotherapist, at the end of the 4-week rehab period under study

CONTACTS AND LOCATIONS:
Overall Officials: Ilaria Baroncini, MD, Principal Investigator — Montecatone Rehabilitation Institute S.p.A.
Locations (1):
- Montecatone Rehabilitation Institute S.p.A., Imola, BO, Italy

IPD SHARING:
Plan to Share IPD: Undecided